CLINICAL TRIAL: NCT05821452
Title: Induction Therapy for Locally Advanced Tumor With Immunotherapy Plus Chemotherapy vs. Chemoradiotherapy for Thoracic Squamous Esophageal Carcinoma
Brief Title: Immunotherapy Plus Chemotherapy vs. Chemoradiotherapy for Thoracic Squamous Esophageal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-ICE Union
Record Dates: First submitted 2023-02-14; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Chemotherapy; Radiation Therapy
Keywords: Immumotherapy plus Chemotherapy; conversion therapy; advanced esophageal squamous cell carcinoma; chemoradiotherapy
MeSH Terms: interventions — camrelizumab; Paclitaxel; Injections; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immumotherapy plus Chemotherapy (Experimental): Paclitaxel: 175mg/m2, intravenous infusion on the first day of each cycle, every 3 weeks for a cycle (Q3W), a total of 3 cycles.
  Cisplatin: 75mg/m2, intravenous infusion on the first day of each cycle, every 3 weeks for a cycle (Q3W), a total of 3 cycles.
  Camrelizumab: 200mg was administered intravenously on the first day of each cycle, every 3 weeks as a cycle (Q3W), for a total of 3 cycles.
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel; Drug: Cisplatin
- chemoradiotherapy (Experimental): Paclitaxel: 175mg/m2, intravenous infusion on the first day of each cycle, every 3 weeks for a cycle (Q3W), a total of two cycles
  Cisplatin: 75mg/m2, intravenous infusion on the first day of each cycle, every 3 weeks for a cycle (Q3W), a total of two cycles
  Radiotherapy: Irradiation mode and dose: three-dimensional conformal or intensity modulated radiotherapy technology was adopted, 41.4Gy, 1.8Gy each time, 5 times a week.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Camrelizumab — 200mgQ3w
  Other Names: pdl1 Inhibitors
  Arms: Immumotherapy plus Chemotherapy
Drug: Paclitaxel — 175mg/m2，D1，Q3w
  Other Names: Paclitaxel For Injection (Albumin Bound)
Drug: Cisplatin — 75mg/m2，D1，Q3w
Radiation: Radiotherapy — 41.4Gy, 1.8Gy each time, 5 times a week
  Other Names: Radiation therapy
  Arms: chemoradiotherapy

SUMMARY:
The investigators conducted a phase II, prospective, two-arm clinical study to explore the efficacy of Camrelizumab combined with chemotherapy versus chemoradiotherapy for conversion therapy of potentially resectable advanced esophageal squamous cell carcinoma. This study will provide more evidence for conversion treatment of initially unresectable locally advanced esophageal squamous cell carcinoma and contribute to the development of treatment guidelines for esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer (EC) has a higher morbidity and mortality rate than most human malignancies. The standard treatment for unresectable locally advanced esophageal squamous cell carcinoma (ESCC) is concurrent chemoradiotherapy, but survival remains limited. Carrilizumab combined with chemotherapy has been shown to have an excellent pathological remission rate in the treatment of advanced esophageal cancer and locally advanced esophageal cancer. Here, the investigators conducted a phase II, prospective, two-arm clinical study to explore the efficacy of Camrelizumab combined with chemotherapy versus chemoradiotherapy for conversion therapy in potentially resectable advanced esophageal squamous cell carcinoma. All participants meeting the inclusion criteria will be registered after signing the informed consent form. Patients with thoracic esophageal cancer with clinical staging of T4a and T4b or at least one group of lymph nodes likely to invade surrounding organs or with concomitant enlarged lymph nodes unresectable will be included in the study. According to the study plan, patients who completed two cycles of chemotherapy combined with Camrelizumab induction or concurrent chemoradiotherapy were randomly assigned to receive radical surgery after being assessed as operable. The primary endpoint was R0 removal rate in patients undergoing surgery after treatment. Secondary endpoints were major pathological response (MPR) rate, overall survival (OS), progression-free survival (PFS), and adverse events. This study will provide more evidence for the conversion treatment of initially unresectable locally advanced esophageal squamous cell carcinoma and contribute to the development of treatment guidelines for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically-confirmed squamous cell carcinoma
* primary lesions located in the thoracic esophagus
* clinical stage cT4 or at least one group of lymph nodes invade the surrounding organs and unresectable lymph nodes
* having not received neoadjuvant therapy
* 18-75 years
* ECOG performance status of 0 or 1
* no prior chemotherapy, radiotherapy, or immunotherapy for any cancers
* adequate organ function
* expectation of R0 resection
* provision of written informed consent.

Exclusion Criteria:

* corticosteroid treatment (equivalent to prednisone >10 mg/day) within 14 days before the first day of the drug administration
* acquired immunodeficiency syndrome or active hepatitis B (DNA ≥ 104 copies/ml) or C (RNA ≥ 103 copies/ml) viral infections
* history of pneumonitis or interstitial lung disease with clinical evidence, such as interstitial pneumonia and pulmonary fibrosis features on baseline CT scans
* known or concurrent bleeding disorders or other uncontrolled diseases contraindicating surgical treatment
* physical examination or clinical trial findings that can interfere with the results or put the patient at increased risk for treatment complications
* comorbidities, including chronic pulmonary disease, poorly controlled hypertension, unstable angina, myocardial infarction within 6 months, and unstable mental disorders requiring therapy
* allergy to drugs used in the study
* participation in other clinical trials within 30 days before enrollment
* ineligibility for participation based on the decision of investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2024-05-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
R0 removal rate | up to 3 months
  R0 removal rate in patients undergoing surgery after treatment
MPR rate | up to 4 months
  major pathological response rate

SECONDARY OUTCOMES:
OS | 12 months
  overall survival
PFS | 12 months
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, Prof, Study Chair — Key Laboratory of Cardio-Thoracic Surgery, Fujian Medical University, Fujian Province University, Fu
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No
Clinical trial registration, unbiased reporting of results and sharing of raw data

REFERENCES:
- [Derived] Chen M, Huang Y, Zhang S, Zheng Y, Zeng T, Chen C, Zheng B. Camrelizumab in combination with chemotherapy versus concurrent chemoradiotherapy for the conversion of locally advanced unresectable oesophageal squamous carcinoma: protocol for a two-arm, open-label phase II trial. BMJ Open. 2024 Feb 28;14(2):e075421. doi: 10.1136/bmjopen-2023-075421. PMID 38418234